CLINICAL TRIAL: NCT06534970
Title: Development, Validation and Clinical Application of a Method for Quantitative 3D Assessment of Facial Symmetry After Facial Reconstruction Using Three-dimensional Stereophotogrammetry
Brief Title: Assessment of Facial Symmetry After Facial Reconstruction Using Three-dimensional Stereophotogrammetry
Acronym: SymFACE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Fondation des Gueules Cassées (Unknown)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0384; ID RCB (Other: 2023-A02406-39)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Facial Reconstruction
Keywords: Three-dimensional stereophotogrammetry; Facial symmetry
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Facial reconstruction patients: Reconstruction of the lower or middle third of the face using a pedicled flap or microanastomosed free flap following excision of a benign or malignant tumor of the oral cavity or face, osteonecrosis of the jaws, or traumatic loss of facial substance
  Interventions: Device: Three-dimensional stereophotogrammetry; Other: Questionnaires

INTERVENTIONS:
Device: Three-dimensional stereophotogrammetry — Three stereoscopic photographs
Other: Questionnaires — * SF-36 quality of life scale for general health inquiry
  * Rosenberg Self-Esteem Scale
  * Self-perception scale

SUMMARY:
Facial reconstruction follows removal of a malignant or benign tumor of the oral cavity or face, complex facial trauma, or resection of osteonecrosis of the jaws. It's a challenge that aims to restore not only the functions of the face, but also its aesthetics, which is just as crucial. A poor aesthetic result after facial reconstruction has a serious impact on patient's lives. To develop more personalized surgery, and to anticipate and correct poor results in the future, it is essential to better understand the factors associated with poor aesthetic results in this type of surgery, as well as their impact on the patient's life.

This means correctly assessing the aesthetic outcome of this surgery. Today, however, aesthetic evaluation criteria remain inadequate. A number of criteria are involved in facial attractiveness, and facial symmetry is a key factor. It is generally accepted that severe facial asymmetries considerably diminish facial attractiveness. Currently, aesthetic evaluation criteria (particularly symmetry) are based primarily on the subjective perception of the surgeon or patient. However, there is a need to be able to measure facial symmetry objectively.

Methods for assessing symmetry rely on the placement of anatomical landmarks and the calculation of Euclidean distance, which involves locating homologous landmarks on each side of the face and comparing the length ratios of all possible lines connecting the landmarks on each side. However, these techniques are based on measurements often on two-dimensional (2D) photographs and do not take into account the three-dimensional nature of the face. Methods for three-dimensional analysis of facial symmetry have been developed based on three-dimensional CT reconstructions. However, this technique implies the use of an irradiating imaging technique, not systematically indicated at a distance from surgery.

This study aims to validate a method for analyzing facial symmetry using three-dimensional stereophotogrammetry, to identify risk factors for facial asymmetry in patients who have undergone facial reconstruction, and to assess the impact of facial asymmetry on patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older,
* Patient having given non-opposition for participation in this study,
* Reconstruction of the lower or middle third of the face by pedicled flap or microanastomosed free flap following excision of a benign or malignant tumor of the oral cavity or face, osteonecrosis of the jaws, loss of facial traumatic substance,
* Surgery and routine follow-up performed in the 3 departments (maxillofacial surgery, ENT, plastic and reconstructive surgery) of the PROMOD cluster at Marseille's CHU Conception

Exclusion Criteria:

* History of reconstruction of the lower or middle third of the face other than that being evaluated at one year for this study,
* Subjects covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship, patients deprived of their liberty, pregnant or breast-feeding women),
* Persons who cannot read and understand the French language well enough to be able to give their non-opposition to participating in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent facial reconstruction, returning for consultation 1 year post-surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between root mean square deviation (RMSE) score and surgeon's assessment score | Day 1

SECONDARY OUTCOMES:
Intraclass Correlation Coefficient to assess intra-operator reproducibility | Day 1
Intraclass Correlation Coefficient to assess inter-operator reproducibility | Day 1
Demographic factors associated with objective facial asymmetry one year after facial reconstruction surgery | Day 1
Clinical factors associated with objective facial asymmetry one year after facial reconstruction surgery | Day 1
Therapeutic factors associated with objective facial asymmetry one year after facial reconstruction surgery | Day 1
Relationship between objective measurement of facial asymmetry and the patient's subjective assessment of perception (satisfaction and body image) | Day 1
  The patient perception score is assessed by a scale constructed by the investigative team.
Relationship between objective measurement of facial asymmetry and the patient's quality of life | Day 1
  The patient quality of life score is assessed by the French-validated SF-36 quality of life scale for general health inquiry" (36 items).
Relationship between objective measurement of facial asymmetry and patient self-esteem | Day 1
  The patient self-esteem score is assessed by the French-validated Rosenberg self-esteem scale (10 items).

CONTACTS AND LOCATIONS:
Overall Officials: CREMIEUX François, Study Director — AP-HM
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided